CLINICAL TRIAL: NCT03564717
Title: Evaluation of Segmented Versus Full Arch Three Dimensionally Printed Transfer Tray for Orthodontic Indirect Bonding: Randomized Controlled Trial
Brief Title: Evaluation of Segmented Versus Full Arch Three Dimensionally Printed Transfer Tray for Orthodontic Indirect Bonding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Alaa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEBD-CU-2018-04-17
Record Dates: First submitted 2018-06-08; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Inaccurate Transfer and Bond Failure of Conventional Indirect Bonding Tray; Accuracy of Bracket Transfer and Bond Failure Rate of Full Arch and Segmented Digitally Printed Trays

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Segmented Three dimensionally printed transfer tray (Experimental)
  Interventions: Other: Segmented three dimensionally printed transfer tray
- Full arch three dimensionally printed transfer tray (No Intervention)

INTERVENTIONS:
Other: Segmented three dimensionally printed transfer tray — Segmented indirect bonding transfer tray
  Arms: Segmented Three dimensionally printed transfer tray

SUMMARY:
This study is conducted to overcome the problems of conventional indirect bonding technique, through investigating accuracy of two novel three dimensionally digitally printed indirect bonding transfer trays (full arch & segmented) in terms of accuracy of transferring brackets, rate of immediate bond failure and chair side time.

DETAILED DESCRIPTION:
Fourteen patients (7 in each group) with mild to moderate crowding, requiring orthodontic treatment with full set of permanent teeth including second molars, will be selected for this study. A total of 196 brackets will be used (98 Full Arch Tray and 98 Segment Arch Tray). The same bracket type and bonding material will used in both groups. The accuracy of bracket transfer will be measured by 3 Shape Ortho planner software (Bracket Placement Module), rate of bond failure by counting number of debonded brackets upon tray removal & chair side time by using digital watch.

ELIGIBILITY:
Inclusion Criteria:

1. Patients seeking fixed orthodontic treatment with full set of permanent teeth including second molars.
2. No sex predilection.
3. Mild to moderate crowding cases (4-6 mm).

Exclusion Criteria:

1. Severely rotated teeth
2. Enamel hypoplasia or hypocalcification.
3. Systemic disease that contraindicates orthodontic treatment.
4. Presence of deep carious lesions or large restorations.
5. No or poor patient's compliance & bad oral hygiene.
6. Psychological problems.

Ages: 16 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of 3D printed full arch &segmented transfer tray. | immediate
  Using Digital Measurements on 3shape software in mm- degrees

SECONDARY OUTCOMES:
Chairside Time | immediate
  Digital stopwatch in seconds
Immediate Bond Failure | immediate
  Counting number of brackets or tubes failed immediately after bonding

IPD SHARING:
Plan to Share IPD: Undecided